CLINICAL TRIAL: NCT05186467
Title: Comparing the Analgesic Effect of Intraperitoneal and Intravenous Magnesium Sulphate in Diagnostic Gynecological Laparoscopy
Brief Title: Pain After Laparoscopy Results From the Incision, Manipulation of the Abdominal Organs, and Retained CO2(Back Pain)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fouad Soliman, Lecturer of Anesthesia and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2007
Record Dates: First submitted 2021-12-29; First posted 2022-01-11 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Post Operative Pain, Acute
Keywords: mgso4,laparoscopy ,intraperitoneal
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraperitoneal magnesium sulfate (IP) group (Active Comparator): They will receive 100 ml normal saline infused over 10 min immediately before the induction of anesthesia and then continuous infusion of 500 ml normal saline intraoperatively then an intraperitoneal wash of 100 ml normal saline containing 30 mg/kg MgSO4 at the end of laparoscopy.
  Interventions: Drug: intraperitoneal Magnesium sulfate
- Intravenous magnesium sulfate (IV) group (Active Comparator): They will receive 100 ml normal saline containing MgSO4 30 mg/kg infused over 10 min immediately before the induction of anesthesia and then continuous infusion of 500 ml normal saline containing MgSO4 (8mg/kg) intraoperatively then intraperitoneal wash using 100 ml normal saline at the end of laparoscopy.
  Interventions: Drug: intravenous magnesium sulfate

INTERVENTIONS:
Drug: intraperitoneal Magnesium sulfate — Intraperitoneal (IP) group will receive 100 ml normal saline infused over 10 min immediately before the induction of anesthesia and then continuous infusion of 500 ml normal saline intraoperatively then intraperitoneal wash of 100 ml normal saline containing 30 mg/kg MgSO4 at the end of laparoscopy.
  Arms: Intraperitoneal magnesium sulfate (IP) group
Drug: intravenous magnesium sulfate — Intravenous (IV) group will receive 100 ml normal saline containing MgSO4 30 mg/kg infused over 10 min immediately before the induction of anesthesia and then continuous infusion of 500 ml normal saline containing MgSO4 (8mg/kg) intraoperatively then intraperitoneal wash using 100 ml normal saline at the end of laparoscopy.
  Arms: Intravenous magnesium sulfate (IV) group

SUMMARY:
Postoperative pain after laparoscopy may be localized pain resulting from incision due to many (two or three) punctures (somatic pain) or due to manipulation of the intra-abdominal organs as ovaries, uterus, omentum, and intestine (visceral pain) or shoulder and back pain caused by retained CO2 in the peritoneal cavity with its irritation effect on the diaphragm.Patients will be divided into two groups:

Intraperitoneal (IP) group (20 patients):They will receive 100 ml normal saline infused over 10 min immediately before the induction of anesthesia and then continuous infusion of 500 ml normal saline intraoperatively then intraperitoneal wash of 100 ml normal saline containing 30 mg/kg MgSO4 at the end of laparoscopy.

Intravenous (IV) group (20 patients):They will receive 100 ml normal saline containing MgSO4 30 mg/kg infused over 10 min immediately before the induction of anesthesia and then continuous infusion of 500 ml normal saline containing MgSO4 (8mg/kg) intraoperatively then intraperitoneal wash using 100 ml normal saline at the end of laparoscopy

ELIGIBILITY:
Inclusion Criteria:

20-44 years old females, (ASA) class I-II

Exclusion Criteria:

* Patient refusal
* Allergy to MgSO4
* Atrio-ventricular conduction abnormalities
* Drug abuse
* Renal or hepatic or cardiovascular dysfunction
* Prior long-term treatment with calcium channel blockers or magnesium

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-02-02 (Estimated); Study Completion 2022-02-05 (Estimated)

PRIMARY OUTCOMES:
Time for first dose of rescue analgesia | 8 hours
  1st time to feel pain
total analgesic doses | 8 hours
  total (ketorolac) analgesic consumption

SECONDARY OUTCOMES:
post operative pain | 8 hours
  The visual analog scale(0-10 with 0 is no pain and 10 is maximum intolerable pain)
sedation | 8 hours
  4 points sedation scale: 0= alert and conscious
  1 =quietly awake 2= asleep but easily arousable 3= deep sleep
adverse events | 8 hours
  side effects
serum mgso4 level | 2 hours
  serum level of mgso4 at end of operation and after 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Soliman, Principal Investigator — Sohag University
Locations (1):
- Fouad Soliman, Sohag, Egypt